CLINICAL TRIAL: NCT00929097
Title: Implementation of Guidelines on Hereditary or Familial Colorectal Cancer Risk Calculation and Risk Communication
Brief Title: Implementation of Guidelines on Hereditary or Familial Colorectal Cancer
Acronym: RISCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Collaborators: Cardiff University (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Comprehensive Cancer Centres (Unknown)
Responsible Party: E.A.R.J. Lohman, Chairman Hospital Board, Radboud University Nijmegen Medical Centre
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZonMw 80-82315-98-09005
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Neoplasms, Hereditary Nonpolyposis
Keywords: Colorectal Neoplasms, (Hereditary Nonpolyposis); Guideline; Health Plan Implementation; Decision Support Techniques; Risk assessment; Familial colorectal cancer risk; Risk assessment tool
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation aids (Experimental)
  Interventions: Other: Implementation aids
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Implementation aids — * Patients and clinicians have access to a website with information on familial colorectal cancer risk; a risk assessment tool and decision aids
  * Clinicians receive the guidelines and a risk communication tool, as well as education
  Arms: Implementation aids
Other: Control — Dissemination of guidelines
  Arms: Control

SUMMARY:
The aim of this study is to improve clinicians' calculation, interpretation and communication of familial colorectal cancer risk, as well as patients' risk perception and uptake of referral for genetic counselling or for surveillance by colonoscopy for their relatives at risk.

DETAILED DESCRIPTION:
Regular colonoscopy is effective in reducing morbidity and mortality due to colorectal cancer (CRC) in patients at increased familial CRC risk. Currently, the majority of these at-risk individuals are not properly referred for increased surveillance by colonoscopy or genetic counselling. In 2008, a national multidisciplinary evidence-based guideline on familial and hereditary CRC was launched in the Netherlands. Clinicians have new tasks in familial CRC risk calculation, interpretation and communication. A clustered randomized controlled trial including an effect, process and cost evaluation will be conducted in eighteen Dutch hospitals to determine the most cost effective way to implement these new guidelines.

Surgeons and gastroenterologists in both the intervention group and the control group will receive background information on familial colorectal cancer risk and the guidelines. Patients and clinicians in the intervention group will receive an additional intervention strategy.

The effect evaluation is done by assessing the number of CRC patients for whom correct risk calculation, interpretation and communication is performed, as well as patients' uptake of the recommended follow up policy. The actual exposure to the different elements of the implementation procedure and the experiences of users will be assessed in the process evaluation. The costs of the implementation procedure will be determined by means of a cost evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colorectal cancer before the age of 70
* Diagnosed in one of the participating hospitals
* Able to read and understand Dutch

Exclusion Criteria:

* Previous referral for genetic counseling

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-07 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
The number of colorectal cancer patients following the most optimal follow up program according to the guidelines. | 1 year

SECONDARY OUTCOMES:
The number of patients for whom MSI testing was performed based on the MIPA criteria | 1 year
The number of CRC patients for whom a correct familial CRC risk is calculated by clinicians (as compared to formally calculated risks) | 1 year
The number of CRC patients for whom a calculated familial CRC risk is correctly interpreted by clinicians | 1 year
The number of CRC patients with whom a calculated familial CRC risk and/or follow up policy is communicated by clinicians | 1 year
Patients' uptake of the follow up policy | 1 year
Actual exposure to the different elements of the implementation strategy | 1 year
Experiences of clinicians and patients with the different elements of the implementation strategy | 1 year
Costs of the implementation procedure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicoline Hoogerbrugge, MD, PhD, Principal Investigator — Radboud University Medical Center; Rosella PMG Hermens, PhD, Principal Investigator — Radboud University Medical Center

REFERENCES:
- [Derived] Dekker N, Hermens RP, Nagengast FM, van Zelst-Stams WA, Hoogerbrugge N; RISCO study group. Familial colorectal cancer risk assessment needs improvement for more effective cancer prevention in relatives. Colorectal Dis. 2013 Apr;15(4):e175-85; discussion p.e185. doi: 10.1111/codi.12117. PMID 23451840
- [Derived] Dekker N, Hermens RP, Elwyn G, van der Weijden T, Nagengast FM, van Duijvendijk P, Salemink S, Adang E, van Krieken JH, Ligtenberg MJ, Hoogerbrugge N. Improving calculation, interpretation and communication of familial colorectal cancer risk: protocol for a randomized controlled trial. Implement Sci. 2010 Jan 28;5:6. doi: 10.1186/1748-5908-5-6. PMID 20181032